CLINICAL TRIAL: NCT03999034
Title: Evaluation of a New Screening Test of Cognitive Impairment Among Multiple Sclerosis Patients
Brief Title: XO as a Screening Test of Cognitive Impairment in Multiple Sclerosis
Acronym: XO-SEP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Merck Santé SAS (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RNI 2019 CLAVELOU (XO et SEP); 2019-A00801-56 (Other: ANSM)
Record Dates: First submitted 2019-06-24; First posted 2019-06-26 (Actual); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Sclerosis, Multiple; Cognitive Dysfunction
Keywords: screening test; XO test
MeSH Terms: conditions — Multiple Sclerosis; Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: Every patients and healthy controls will fill in all the tests and questionnaires
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients (Experimental): experimental, cognitive test, no treatment investigated. 140 patients (90 relasping remitting and 50 progressive multiple sclerosis)
  Interventions: Diagnostic Test: questionnaire completion
- Healthy controls (Experimental): experimental, cognitive test, no treatment investigated. 400 healthy controls divided into 20 groups, due to gender, age (5 classes: 18-33, 34-43, 44-54, 55-64, and more than 65 years old), and level of education (graduated or not).
  Interventions: Diagnostic Test: questionnaire completion

INTERVENTIONS:
Diagnostic Test: questionnaire completion — Every patient (140) and healthy control (400) will fill in all the tests and questionnaires, except FSS, in a random order during a single appointment. The FSS will be fill in by patients only. All 400 healthy controls will be divided in 20 groups of 20 people, according to gender, age (5 classes: 18-33, 34-43, 44-54, 55-64, and more than 65 years old), and level of education (graduated or not). 60 of them will pass the XO test at the beginning and again at the end of the consult to investigate the test-retest effect.

SUMMARY:
Even at the disease onset, about 70% of patients with multiple sclerosis (MS) suffer from cognitive impairment that impacts quality of life. Currently, some speed processing tests are used, such as SDMT ( symbol digit modalities test ), CSCT (information treatment speed evaluation) and WAIS-IV (Weschler Adult Intelligence Scale ). Their inconvenient are the improvement of scores in test-retest, and some difficulties doing the tests due to motor or visual impairment that might be reported. The XO test is fast, cheap and easy to use during medical consult by neurologists. It seems to be correlated to results of speed processing tests, and probably to some executive functions tests too. Asthenia, anxiety, depression and pain are likely to have a negative influence on tests results. Screening every patients with a short test aims to detect patients with cognitive impairment earlier. After a positive screening test, and to better characterize cognitive impairment, they will undergo a neuropsychological test battery. Depending on the alteration, adapted workstation, financial support, technical and human helps will be implemented in order to improve the daily-living of patients.

This study aims to approve the XO as a screening test of cognitive impairment in MS patients. We will study the relationship between XO test, and SDMT, CSCT, WAIS-IV, and also with questionnaires about pain, asthenia (FSS, Fatigue Severity Scale), anxiety and depression (HAD, Hospital Anxiety and Depression ). The XO test will be standardized using a healthy population.

DETAILED DESCRIPTION:
Even at the disease onset, about 70% of patients with multiple sclerosis (MS) suffer from cognitive impairment that impacts quality of life. Currently, some speed processing tests are used, such as SDMT, CSCT and WAIS-IV. Their inconvenient are the improvement of scores in test-retest, and some difficulties doing the tests due to motor or visual impairment that might be reported. The XO test is fast, cheap and easy to use during medical consult by neurologists. It seems to be correlated to results of speed processing tests, and probably to some executive functions tests too. Asthenia, anxiety, depression and pain are likely to have a negative influence on tests results. Screening every patients with a short test aims to detect patients with cognitive impairment earlier. After a positive screening test, and to better characterize cognitive impairment, they will undergo a neuropsychological test battery. Depending on the alteration, adapted workstation, financial support, technical and human helps will be implemented in order to improve the daily-living of patients.

This study aims to approve the XO as a screening test of cognitive impairment in MS patients. We will study the relationship between XO test, and SDMT, CSCT, WAIS-IV, and also with questionnaires about pain, asthenia (FSS), anxiety and depression (HAD). The XO test will be standardized using a healthy population. 140 multiple sclerosis patients (90 relapsing remitting, and 50 progressive) and 400 healthy controls must be recruited.

Multiple sclerosis patients included must :

* Be men or women aged 18 or more
* Be diagnosed with Multiple Sclerosis (MacDonald criteria, 2017)
* Absence of relapse in the previous month
* Be mother-tongue French, or speaking French fluently
* Be covered by French social security

Healthy controls included must :

* Be men or women aged 18 or more
* Suffer from no pathology that might be incompatible with the study

People who can't be included :

* Patients or controls declining participation to the study, or legally protected, pregnant or breastfeeding women
* Patients suffering from another neurological disease, psychiatric disorder, or developmental abnormalities that were diagnosed before multiple sclerosis
* Patients with cranial trauma, relapse that ended less than 1 month before, or depression in the last 3 months
* Patients with severe motor or visual disabilities There are 4 centers. This is a prospective cohort study, in which data will be collected during a single appointment.

The score obtained doing XO test is the dependent variable that will be compared to the variables due to speed processing and executive functions tests. Test-retest of XO test will also be assessed. The percentage of wrong answers doing XO test will be investigated.

The study is going to last 18 months. Every patient (140) and healthy control (400) will fill in all the tests and questionnaires, except FSS (fatigue severity scale), in a random order during a single appointment. The FSS will be filled in by patients only. All 400 healthy controls will be divided in 20 groups of 20 people, due to gender, age (5 classes: 18-33, 34-43, 44-54, 55-64, and more than 65 years old), and level of education (graduated or not). 60 of them will undergo the XO test at the beginning and again at the end of the appointment to investigate the test-retest effect.

ELIGIBILITY:
Inclusion criteria :

* Multiple sclerosis patients included must :
* Be men or women aged 18 or more
* Be diagnosed Multiple Sclerosis (MacDonald criteria, 2017)
* No relapse in the previous month
* Be mother-tongue French, or speaking French fluently
* Be covered by French social security

Healthy controls included must :

* Be men or women aged 18 or more
* Suffer from no pathology that might be incompatible with the study

Exclusion criteria :

* - Patients or controls declining participation to the study, or legally protected, pregnant or breastfeeding women
* Patients suffering from another neurological disease, psychiatric disorder, or developmental abnormalities that were diagnosed before multiple sclerosis
* Patients with cranial trauma, relapse that ended less than 1 month before, or depression less than 3 months
* Patients with severe motor or visual disabilities

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 540 (Estimated)
Dates: Start 2019-07-08 (Actual); Primary Completion 2020-09-08 (Estimated); Study Completion 2020-10-08 (Estimated)

PRIMARY OUTCOMES:
Score of XO test | Day 0
  The score obtained doing XO test is the dependent variable that will be compared to the variables due to speed processing and executive functions tests. Test-retest of XO test will be also assessed. The percentage of wrong answers doing XO test will be investigated.

SECONDARY OUTCOMES:
Score of anxiety | Day 0
  Every patients and healthy control will fill in the HAD questionnaire, exploring both anxiety and depression. It is composed of 7 questions ranged from 0 to 3. The test score is ranged from 0 to 21. Higher values are correlated to worse outcome.The score of anxiety is an independent variable that will be compare to score of XO test.
Score of depression | Day 0
  Every patients and healthy control will fill in the HAD questionnaire, exploring both anxiety and depression. It is composed of 7 questions ranged from 0 to 3. The test score is ranged from 0 to 21. Higher values are correlated to worse outcome.The score of depression is an independent variable that will be compare to score of XO test.
Score of asthenia | Day 0
  Every patients and healthy control will fill in the FSS (fatigue severity scale) questionnaire, exploring asthenia in Multiple Sclerosis patients. It is composed of 9 questions ranged from 1 to 7. The test score is ranged from 9 to 63. Higher values are correlated to worse outcome. The score of asthenia is an independent variable that will be compared to score of XO test.
Score of pain | Day 0
  Every patients and healthy control will fill in a pain questionnaire, exploring both cephalalgia, nociceptive and neuropathic pain. It is composed of 22 questions. Some questions must be answered by "yes" or "no". Some other questions are using a visual analogue pain scale from 0 to 10, where 10 is the worse outcome. Some questions need to write the topography of the pain, and the treatment used. Every answer to the questionnaire of pain is an independent variable that will be compare to score of XO test.

CONTACTS AND LOCATIONS:
Overall Officials: Pierre CLAVELOU, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France